CLINICAL TRIAL: NCT06584721
Title: Comparison of Short Foot Exercises and Anti-pronation Taping on Low Back Pain Associated With Hyper Pronation of Foot
Brief Title: Short Foot Exercises and Anti-pronation Taping on Low Back Pain Associated With Hyper Pronation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01876 Sunbal Fatima
Record Dates: First submitted 2024-09-02; First posted 2024-09-05 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain
Keywords: Short foot exercises; Foot hyper-pronation; low back pain; Anti-pronation Taping
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-pronation taping (Low dye taping) + Conventional therapy (Active Comparator): Anti-pronation taping and conventional
  Interventions: Other: Anti-pronation taping (Low dye taping) + Conventional therapy
- Short Foot Exercises + Conventional Study (Other): Short foot exercises + Conventional therapy
  Interventions: Other: Short Foot Exercises + Conventional PT

INTERVENTIONS:
Other: Anti-pronation taping (Low dye taping) + Conventional therapy — They would be receiving treatment as follow:
  Anti-pronation taping (Low dye taping) Applied on alternate days. 3 days / week for 4 weeks.
  Conventional Therapy includes 1. Tens biphasic mode, 90Hz, 100ms pulse width for 20 mins 2. William flexion exercises (5repsx1set). 3. Lower limb stretching exercises (3repsxset1, 10sec hold) 3sessions/ week.
  Arms: Anti-pronation taping (Low dye taping) + Conventional therapy
Other: Short Foot Exercises + Conventional PT — They would be receiving treatment as follow:
  Short foot exercises are used to reduce the foot pronation: Frequency: 30 reps x 1 set, 30 sec hold and 10 sec relaxation for 4 weeks. 3 session/ week).
  Short foot Exercises includes a four-week plan, 1- Shortening of foot in Anterior-posterior direction, 2- Increase medial longitudinal arch, 3- Balanced loading in standing, 4- Approximating Head of first, second meta-tarsal and calcaneus with patient in standing (single leg).
  Conventional therapy includes 1. Tens biphasic mode, 90Hz, 100ms pulse width for 20 mins 2. William flexion exercises (5repsx1set). 3. Lower limb stretching exercises (3repsx1set, 10sec hold) 3sessions/ week.
  Arms: Short Foot Exercises + Conventional Study

SUMMARY:
The aim of this randomized clinical trial is to find the comparison of Short foot exercises and anti-pronation taping on low back pain associated with hyper pronation on reducing back pain improving range of motion of foot, back and foot posture.

DETAILED DESCRIPTION:
Low back pain is a musculoskeletal symptom which occur in all ages during life time with acute episode or chronic condition. Total of 619 million people are living with low back pain worldwide. Low back pain is the musculoskeletal condition that involves pain in region below costal margin and above inferior gluteal fold, along with pain there is also stiffness, limitation of range of motion, aggravated by movement and affected ability to perform daily life activities. Frequency and severity of low back pain are related to spinal loading that increase the strain on lumbar spine, these loads shift from foot (during heel strike) to leg and ultimately to the back.

Abnormal mechanical loading of lumbar spine due to poor postural control or muscular weakness is considered as risk factor for low back pain. The ability of ankle complex to provide stabilization and mobilization depends upon plantar pressure distribution. In particular, pronated foot causes internal rotation of tibia along with internal rotation of hip that cause femoral ante-version and increase in lumbar lordosis and deteriorate lumbopelvic alignment resulting in low back pain Short foot exercise (SFE) is considered more effective in terms of postural balance and excessive pronation. SFE is a widely used intervention that has been developed recently to improve ankle proprioception and global movement pattern, so as to elevate and support the medial longitudinal arch of the foot and to improve dynamic standing balance Anti-pronation taping is a technique that stimulate underlying sensory receptor either through the surface contact or stretch of skin that causes the sensory input to central nervous system to be altered hence it ultimately influences the execution and perception of movement. Low dye taping is effective in correcting over-pronated foot and also increase navicular height along with increase in reactive strength index. low dye taping not only improve arch height but also improves muscular activity The rationale for the use of these techniques is to compare the effect of short foot exercises and anti-pronation taping on low back pain associated with hyper-pronated foot and also on range of motion of foot and back along with the foot posture.

ELIGIBILITY:
Inclusion Criteria

* Both gender
* Age 25 to 45 years
* Foot hyper pronation (FPI ≥ +6)
* low back pain > 3months (Pain, muscle stiffness, and muscle tension between lower costal margin and inferior gluteal fold)
* Low back pain with NPRS ≥ 3

Exclusion Criteria:

* Acute trauma or fracture of foot/ back (last 3 months)
* leg length discrepancy >5mm
* Diagnosed with Spondylolisthesis, spondylitis
* Diagnosed with Lumbar radiculopathy, stenosis, fibromyalgia, plantar fasciitis
* Recent History of fall < 3months
* Congenital hyper-pronation of foot
* Pregnancy

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-08-27 (Estimated); Study Completion 2025-08-27 (Estimated)

PRIMARY OUTCOMES:
Range of motion (Goniometer) | 4 weeks
  It is a tool used to measure the range of motion of joint (0-180). Record the starting measurement, remove the goniometer, and allow the patient to move the joint through the available range of motion. Replace and realign the goniometer. Read and record the measurement.
Numeric Pain Rating Scale NPRS | 4 weeks
  The NPRS is an eleven-point pain impression scale: the patient rates pain from 0 (no aggravation) to 10 (most exceedingly terrible possible pain). Numeric Pain Rating Scale (NPRS), which was used to survey respondents' impression of the degree of pain that they felt. NPRS has been utilized in different examinations for low back pain.
Foot Posture Index | 4 weeks
  It is a tool which provides quantitative data about foot posture. It has total six items. Talar head palpation, observation of curves above and below the lateral malleolus, a bulge in the region of the talonavicular joint, eversion and inversion of the calcaneus, congruence of the medial longitudinal arch, adduction and abduction of the forefoot in relation to the rear foot. Total score between (- 12 and + 12). (0 and + 5 normal feet) ;( + 6 to + 9 pronated feet) ;( ≥ + 10 highly pronated feet) ;( - 1 to - 4 supinated feet); - 5 to - 12 indicate highly supinated.
Oswestry Disability Index | 4 weeks
  The ODQ scale was utilized to quantify the limitations in regular daily life activities. It depends on 10 segments with six levels each, evaluating the restriction of different activities of day to day living. The qualities range from 0 (the best wellbeing state) to 100 (the most worsening wellbeing state). For each segment of the poll, the absolute plausible score is 5.

CONTACTS AND LOCATIONS:
Overall Officials: Kinza Anwar, MS, Principal Investigator — Riphah International University
Locations (1):
- Rawal Surgical Hospital, Nawababad, Wah Cantt, Wāh, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No